CLINICAL TRIAL: NCT01878084
Title: Phase I/II Trial of Alveolar Bone Engineering Using Bioactive Glass (Sol-Gel) Immediately After Premolar Extraction in Patients Requiring Orthodontic Treatment
Brief Title: Bioactive Glass (Sol-gel) for Alveolar Bone Regeneration After Surgical Extraction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Collaborators: Lehigh University (Other)
Responsible Party: Principal Investigator, Prof. Mona K. Marei, professor/head of tissue engineering laboratories, faculty of dentistry, Alexandria University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BIOGLASS-STDF#116
Record Dates: First submitted 2013-06-10; First posted 2013-06-14 (Estimated); Results first posted 2020-02-18 (Actual); Last update posted 2020-02-18 (Actual); Status verified 2020-02

CONDITIONS: Bone Loss; Vertical Alveolar Bone Loss; Horizontal Alveolar Bone Loss
Keywords: Tissue regeneration; sol gel bioglass; alveolar ridge preservation; children; Egyptian; class II orthodontic cases
MeSH Terms: conditions — Bone Diseases, Metabolic

STUDY DESIGN:
Intervention Model Description: This study represents a split-mouth study where the right or left/ upper or lower premolar could be assigned to either the control group (socket left empty) or test group (socket filled with bioactive glass (sol-gel)
  The extraction sockets will be allocated either to the control : Extraction socket will be left empty
  or
  Test: Extraction socket will be augmented using bioactive glass (sol-gel)
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- all study participants (Other): This study represents a split-mouth study where the right or left/ upper or lower premolar could be assigned to either the control group (socket left empty) or test group (socket filled with bioactive glass (sol-gel)
  The extraction sockets will be allocated either to the control : Extraction socket will be left empty
  or
  Test: Extraction socket will be augmented using bioactive glass (sol-gel)
  Interventions: Other: bioactive glass (sol-gel); Other: empty extraction socket

INTERVENTIONS:
Other: bioactive glass (sol-gel) — Extraction sockets will be augmented using bioactive glass (sol-gel)
  Other Names: Tailored Amorphous Multiscale Porous (TAMP) scaffold
Other: empty extraction socket — Extraction socket will be left empty

SUMMARY:
The purpose of the present research is to evaluate the effect of bioactive glass in bone regeneration immediately following extraction of mandibular and maxillary premolars.The hypothesis of the study assumes that this treatment would promote the healing of the extraction socket while preserving both the height and width of the bone. Furthermore, it would allow more effective tooth movement during orthodontic treatment.

DETAILED DESCRIPTION:
Bioactive glass has long been known as a bone graft substitute capable of bone augmentation. The current proposal introduces a newly tailored bioactive glass scaffold with multi-scale porosity prepared using the sol-gel technique to regenerate bone in extraction sockets with the aim of preserving the alveolar ridge. This novel material has the potential to enhance angiogenesis and osteogenesis thereby preserving the overall height and width of the alveolar bone by regenerating new bone that closely mimics the adjacent healthy one. Thirty patients requiring myofunctional therapy including premolar extraction as part of a two stage orthodontic treatment (class II division I) will be enrolled in this phase I/II clinical study. Patients will undergo extraction of their maxillary and mandibular premolar teeth. This will serve as a split-mouth study where on one side the extraction sockets will be left empty while on the other side they will receive the bioactive glass as a bone graft substitute. Clinical and radiographic assessment of healing will be performed at the following time intervals; 1,2,4,12,24 weeks. Clinical criteria will include scoring for pain, inflammation, and occurrence of any post-operative complications using a well-defined scoring system. Radiographic assessment will monitor the changes in crestal bone height and bone mineral density. Computed tomographic scans will also be taken preoperatively and at 6 months for each patient for 3D assessment of bone changes. A core biopsy will also be taken after informed consent at the 6 months time-point to evaluate the quality and quantity of new bone formed.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have good oral hygiene (confirmed by OHI-S)
* Patients who had voluntarily agreed on signing an informed consent including the duration and all the steps of the trial
* Patients who are indicated for the administration of the type of local anesthesia used in the trial
* Patients who need myofunctional therapy including premolar extraction as part of two stage treatment (class II division I)
* Patients indicated for premolar extraction as a normal step in the treatment plan not intentionally for the experiment.
* Patients who had undergone x- rays on the premolar teeth showing root form and the shape of the socket prior to extraction

Exclusion Criteria:

* Patients with history of bleeding disorders which will hinder the normal healing process of the needed sockets for the trial
* Patients with history of allergy to foreign bodies , i.e. susceptible to reactions from Bioglass
* Patients with history of hypertension and diabetes , rendering them not indicated for administration of the recommended type of local anesthesia nor even for extraction
* Patients having HCV , HBV , HIV or other infectious diseases to make sure of the safety of the research team and the participants from probable infection .
* Mentally retarded patients who are not able to understand the steps of the trial Patients with systemic diseases or febrile illness making them unable to follow the appointments arranged
* Patients who simultaneously participate in other research studies
* Patients with traumatic surgical extraction

Ages: 9 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 9 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2018-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mona Marei, prof, Principal Investigator — Alexandria University
Locations (1):
- Tissue Engineering Laboratories, Faculty of Dentistry, Alexandria University, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] El Shazley N, Hamdy A, El-Eneen HA, El Backly RM, Saad MM, Essam W, Moussa H, El Tantawi M, Jain H, Marei MK. Bioglass in Alveolar Bone Regeneration in Orthodontic Patients: Randomized Controlled Clinical Trial. JDR Clin Trans Res. 2016 Oct;1(3):244-255. doi: 10.1177/2380084416660672. Epub 2016 Aug 6. PMID 30931746

RESULTS

PARTICIPANT FLOW:
Recruitment Details: participants were recruited from the outpatient clinic of the orthodontic department at the Faculty of Dentistry of Alexandria University From October 2013 to October 2014
Units Other Than Participants: extraction socket
Groups:
- All Study Participants: Bone regeneration utilizing tissue engineering principles and approach via using porous bioactive glass prepared by sol gel technique to properly fill the empty socket after tooth extraction. The target is to preserve the buccal and lingual alveolar plates of the socket regarding width and height, to avoid bone resorption and to stimulate bone regeneration. This novel technique will be evaluated via histological (biopsy), radiographic, and bone density measurements in addition to clinical assessment.
  This study represents a split-mouth study where the right or left/ upper or lower premolar could be assigned to either the control group (socket left empty) or test group (socket filled with bioactive glass (sol-gel)
  The extraction sockets will be allocated either to the control : Extraction socket will be left empty
  or
  Test: Extraction socket will be augmented using bioactive glass (sol-gel)
Period: Overall Study
Arm/Group | All Study Participants
Started | 9; 18 extraction socket
Test(Received TAMP Bioglass) s | 7; 7 extraction socket
Control (Sockets Were Left Empty) | 7; 7 extraction socket
Completed | 7; 14 extraction socket
Not Completed | 2; 4 extraction socket
Not completed — Physician Decision | 2

BASELINE CHARACTERISTICS:
Population: This is a split mouth study design, and so each patient serves as both test and control.
Arm/Group | All Study Participants
Number analyzed (Participants) | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 12 (1.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 2
Race/Ethnicity, Customized [Number; unit: participants]
  Egyptians | 7
Region of Enrollment [Number; unit: participants]
  Egypt | 7

OUTCOME MEASURES:

1. Primary Outcome: Change in Alveolar Crestal Bone Height
Description: The primary objective of the study is to determine the effect of using bioactive glass in preservation of alveolar crestal height and width surgical sockets immediately after premolar extraction assessed at baseline, 1,2,4,8,12,24 weeks post-extraction, baseline ,4 and 12 weeks reported. This change was analyzed by subtracting the values of each interval from the baseline values.the positive values indicate that the alveolar crest is coronal to the cemento enaml junction (reference point) , while the negative values indicate that the alveolar crest in apical to the cemento enamel junction (reference point)
Time Frame: assessed at baseline, 1,2,4,8,12,24 weeks post-extraction, baseline,4 and 12 weeks reported.
Population: previously described
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: extraction sockets
Groups:
- All Study Participants: This study represented a split-mouth study where the right or left/ upper or lower premolar was assigned to either the control group (socket left empty) or test group (socket filled with bioactive glass (sol-gel)
  The extraction sockets were allocated either to the control : Extraction socket were left empty
  or
  Test: Extraction socket were augmented using bioactive glass (sol-gel
  bioactive glass (sol-gel): Extraction sockets were augmented using bioactive glass (sol-gel)
Arm/Group | All Study Participants
Number analyzed (Participants) | 7
Number analyzed (extraction sockets) | 14
mm
  baseline control mesial alveolar bone height value | 0.32 (0.76)
  baseline test mesial alveolar bone height value | 0.84 (1.57)
  baseline control distal alveolar bone height value | 1.59 (1.03)
  baseline test distal alveolar bone height value | 0.96 (1.57)
  4 weeks control mesial alveolar bone height value | -0.11 (0.95)
  4 weeks test mesial alveolar bone height value | -0.36 (1.40)
  4 weeks control distal alveolar bone height value | 1 (1.28)
  4 weeks test distal alveolar bone height value | 0.03 (1.76)
  12 weeks control mesial alveolar bone height value | -0.13 (0.25)
  12 weeks test mesial alveolar bone height value | 0.08 (1.09)
  12 weeks control distal alveolar bone height value | 0.33 (0.8)
  12 weeks test distal alveolar bone height value | 0.47 (0.98)

2. Primary Outcome: Bone Mineral Density
Description: The primary objective of the study is to determine the effect of using bioactive glass in inducing alveolar bone regeneration safely and effectively in surgical sockets immediately after premolar extraction assessed at baseline, 1,2,4,8,12,24 weeks post-extraction, baseline,4 and 12 weeks reported.
Time Frame: assessed at baseline, 1,2,4,8,12,24 weeks post-extraction, baseline,4 and 12 weeks reported.
Population: previously described
Measure: Mean (Standard Deviation); unit: percentage of BMD
Units Other Than Participants: extraction sockets
Groups:
- All Study Participants: This study represented a split-mouth study where the right or left/ upper or lower premolar were assigned to either the control group (socket left empty) or test group (socket filled with bioactive glass (sol-gel)
  The extraction sockets were allocated either to the control : Extraction socket were left empty
  or
  Test: Extraction socket were augmented using bioactive glass (sol-gel
Arm/Group | All Study Participants
Number analyzed (Participants) | 7
Number analyzed (extraction sockets) | 14
percentage of BMD
  baseline control coronal bone density value | 38.30 (14.94)
  baseline test coronal bone density value | 42.28 (19.50)
  baseline control middle bone density value | 63.32 (16.20)
  baseline test middle bone density value | 55.92 (17.24)
  baseline control apical bone density value | 75.17 (13.12)
  baseline test apical bone density value | 75.61 (16.72)
  4 weeks control coronal bone density value | 39.54 (17.14)
  4 weeks test coronal bone density value | 40.03 (14.83)
  4 weeks control middle bone density value | 67.29 (18.28)
  4 weeks test middle bone density value | 68.95 (16.94)
  4 weeks control apical bone density value | 76.47 (14.42)
  4 weeks test apical bone density value | 83.98 (13.30)
  12 weeks control coronal bone density value | 47.71 (14.85)
  12 weeks test coronal bone density value | 49.44 (13.92)
  12 weeks control middle bone density value | 66.59 (15.76)
  12 weeks test middle bone density value | 67.14 (11.05)
  12 weeks control apical bone density value | 74.10 (12.08)
  12 weeks test apical bone density value | 76.15 (13.41)

ADVERSE EVENTS:
Description: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed; Since the material used has been previously tested for other bone applications and no adverse events were reported.
Groups:
- All Study Participants: This study represented a split-mouth study where the right or left/ upper or lower premolar were assigned to either the control group (socket left empty) or test group (socket filled with bioactive glass (sol-gel)
  The extraction sockets were allocated either to the control : Extraction socket were left empty
  or
  Test: Extraction socket were augmented using bioactive glass (sol-gel)
Arm/Group | All Study Participants
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes